CLINICAL TRIAL: NCT03546049
Title: Prospective Multi-site Study of Ultrasound-guided Percutaneous Biliary Drainage and Endoscopic Ultrasound-guided Biliary Drainage With Implantation of a Self-expanding Metal Stent in Patients With Malignant, Distal Bile Duct Obstruction
Brief Title: Ultrasound-guided Percutaneous Biliary Drainage Versus Endoscopic Ultrasound-guided Biliary Drainage
Acronym: PUMa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Theresienkrankenhaus und St. Hedwig-Klinik GmbH (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Daniel Schmitz, MD, Medical doctor, assistant medical director, Theresienkrankenhaus und St. Hedwig-Klinik GmbH
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-PUMa-3-12-001
Record Dates: First submitted 2018-03-15; First posted 2018-06-06 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Bile Duct Obstruction, Extrahepatic
Keywords: ultrasound-guided percutaneous transhepatic biliary drainage; endoscopic ultrasound-guided antegrade biliary drainage; endoscopic ultrasound-guided transhepatic biliary drainage; endoscopic ultrasound-guided choledochal biliary drainage; self-expandable metal stent; malignant bile duct obstruction
MeSH Terms: conditions — Cholestasis, Extrahepatic

STUDY DESIGN:
Intervention Model Description: prospective, non-randomized multicenter study (each center performs the intervention which can do best)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-guided percutaneous biliary drainage (Active Comparator): The initial percutaneous transhepatic puncture of the bile duct is performed by ultrasound guidance with a Chiba-needle (0.7 mm). After injection of a radiopaque contrast media into the bile duct system, the malignant extrahepatic bile duct stenosis can be visualized by fluoroscopic guidance (digital remote-controlled fluoroscopy device). Then a 0.018 inch guide wire is introduced and proceeded beyond the tumor stenosis into the duodenum. Next, the Chiba needle is exchanged by a 5 F catheter and the 0.018 inch guide wire is exchanged by a 0.035 inch guide wire. After dilatation of the hepatic access route with bougies up to 12 F, a self-expandable metal stent is introduced. The placement of the metal stent is controlled by endoscopic luminal guidance (gastroscope or duodenoscope).
  Interventions: Procedure: US-guided percutaneous biliary drainage
- EUS-guided biliary drainage (Experimental): The initial transluminal puncture of the bile duct is performed by endoscopic ultrasound guidance (longitudinal echoendoscope) with an 19 G access needle. After injection of a radiopaque contrast media into the bile duct system, the malignant extrahepatic bile duct stenosis can be visualized by fluoroscopic guidance. Then, a 0.035 inch guide wire is introduced into the bile duct. After dilatation of the transluminal access route with a balloon catheter, a self-expandable metal stent is introduced as an antegrade biliary drainage, a transhepatic biliary drainage or a choledochal biliary drainage. The placement of the metal stent is controlled by fluoroscopic and endoscopic luminal guidance.
  Interventions: Procedure: EUS-guided biliary drainage

INTERVENTIONS:
Procedure: US-guided percutaneous biliary drainage — Device: metal stent. The self-expandable metal stent is implanted percutaneously by a transhepatic access route.
  The metal stent is partially covered or non-covered (in cases in which the gallbladder is not removed).
  Length: 6-10 cm. Diameter: 8-10 mm.
  Other Names: WallFlex™ Biliary RX Stents Boston Scientific
  Arms: US-guided percutaneous biliary drainage
Procedure: EUS-guided biliary drainage — Device: metal stent. The transluminal (transgastric, transduodenal or transenteric) implanted self-expandable metal stent is released via echoendoscope.
  The metal stent is partially covered or non-covered (in cases in which the gallbladder is not removed) or mixed covered (one half covered, one half non-covered). The mixed covered stent is used for the transhepatic access.
  Length: 6-10 cm. Diameter: 8-10 mm.
  Other Names: WallFlex™ Biliary RX Stents Boston Scientific
  Arms: EUS-guided biliary drainage

SUMMARY:
Prospective multi-site study of ultrasound-guided percutaneous biliary drainage and endoscopic ultrasound-guided biliary drainage with implantation of a self-expanding metal stent in patients with malignant, distal bile duct obstruction (PUMa-study)

DETAILED DESCRIPTION:
In a recent systematic review and meta-analysis about the efficacy and safety of endoscopic ultrasound-guided biliary drainage (EUBD) in comparison with percutaneous transhepatic biliary drainage (PTBD), there was no difference in technical success between the two procedures, but PTBD was associated with a lower level of clinical success, a higher level of post-procedural adverse events and a higher rate of re-interventions. The authors concluded that EUBD should be favored for biliary drainage when endoscopic retrograde cholangiopancreaticography (ERCP) failed or wasn´t possible to perform due to anatomical reasons.

The hypothesis of this prospective multicenter study is that PTBD wasn´t performed in an appropriate way to compare it adequately with EUBD. The following improvements should be done. First, color Doppler ultrasound-guidance for cannulating the bile duct should be used in PTBD. The transgression of blood vessels with the risk of severe intrahepatic bleedings or hemobilia can be avoided, which are common adverse events in PTBDs when it is performed by fluoroscopic guidance. Second, the access to the bile duct from the left side of the liver should be favored. The access from the right liver side causes more adverse events such as biliary effusion or pneumothorax, as well as more patient discomfort and pain. Third, implantation of the self-expanding metal stent should be performed in the first session as a one-step procedure. This has the advantage that no further re-intervention is necessary after insertion of an external or an external/internal drainage, an outcome which can cause further adverse events such as bile duct leak along the catheter, biliary ascites or catheter dislocation. Fourth, stent release should be performed under endoscopic luminal guidance. In this way, the positioning and the correct expansion of the distal tip of the metal stent can be observed directly in comparison with the stent release which is only controlled by fluoroscopic guidance.

On the other hand, EUBD should be performed in its best manner (special metal stents included) with the three techniques that are usually necessary to perform a successful EUBD: EUS-guided antegrade transpapillary drainage, EUS-guided transhepatic drainage and EUS-guided choledochal drainage.

The study focuses on patients with malignant distal (infra-hilar) bile duct obstruction.

It is presumed that the technical and clinical success rate is equal (non-inferiority) but the adverse event rate, the number of re-interventions and the number of days of hospitalization may differ between the two interventions. An adequate number of cases (106 patients in each intervention, drop outs included) should be recruited to calculate relevant statistical differences.

Furthermore, patients will be followed over six months after the intervention to calculate an estimated survival analysis (with and without palliative chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Inoperable, malignant disease with extrahepatic bile duct obstruction (infra- hilar)
* ERCP was not successful or wasn´t possible due to anatomical reasons (for example status post-gastrectomy)
* At least twofold elevated bilirubin level (> 2mg/dl)
* Histologically verified malignant disease
* Abdominal ultrasound was performed
* Computed tomography or magnetic resonance imaging of the abdomen was performed
* A written consent was given

Exclusion Criteria:

* Relevant blood coagulation disorder (Quick < 50%, Partial thromboplastin time > 50 sec., thrombocytes < 50/nl)
* Extrahepatic cholangiocellular carcinoma (Klatskin tumor) Bismuth II-IV or intrahepatic cholangiocellular carcinoma
* Operable, malignant disease or disease which can be cured by chemotherapy (for example aggressive Non Hodgkin-lymphoma)
* Pregnancy or breastfeeding
* Participation in another trial concerning PTBD or EUBD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Technical success | 1 minute after injection of a radiocontrast agent into the expanded metal stent
  Successful implantation of a self-expanding metal stent to drain the obstructed bile duct, measured by the successful drainage of the radiocontrast agent by the metal stent

SECONDARY OUTCOMES:
Clinical success | 7 days after the intervention
  Decrease of bilirubin level on more than a half of the initial value
Adverse events | Up to 30 days after the intervention
  All adverse events caused by the intervention
Re-interventions | 6 months after successful implantation of the metal stent
  Number of re-interventions (PTBD or EUBD) that are necessary in the follow up (for example due to due stent occlusion or stent migration) after successful stent implantation
Duration of the procedure | The day of the performed procedure (24 h), usually from 10 minutes up to 180 minutes
  Duration of biliary drainage procedure (US-guided percutaneous biliary drainage or EUS-guided biliary drainage) in minutes
Length of hospital stay | The day of the first PTBD or EUBD is counted as day 1 of hospital stay. The day of the discharge from the hospital is counted as the last day of hospital stay. An average 7 to 14 days is estimated.y.
  Length of hospital stay from the day of the first intervention (PTBD or EUBD) to the the day of discharge (days)
Survival time | Follow up of six months
  Time from the day of intervention to the death of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Anja Sander, Dr.M.Sc., Study Director — Institut für Medizinische Biometrie und Informatik Abteilung Medizinische Biometrie, Heidelberg University Hospital
Locations (1):
- Tertiary referral hospital: Theresienkrankenhaus und St. Hedwig Hospital, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharaiha RZ, Khan MA, Kamal F, Tyberg A, Tombazzi CR, Ali B, Tombazzi C, Kahaleh M. Efficacy and safety of EUS-guided biliary drainage in comparison with percutaneous biliary drainage when ERCP fails: a systematic review and meta-analysis. Gastrointest Endosc. 2017 May;85(5):904-914. doi: 10.1016/j.gie.2016.12.023. Epub 2017 Jan 4. PMID 28063840
- [Background] Bapaye A, Dubale N, Aher A. Comparison of endosonography-guided vs. percutaneous biliary stenting when papilla is inaccessible for ERCP. United European Gastroenterol J. 2013 Aug;1(4):285-93. doi: 10.1177/2050640613490928. PMID 24917973
- [Background] Artifon EL, Aparicio D, Paione JB, Lo SK, Bordini A, Rabello C, Otoch JP, Gupta K. Biliary drainage in patients with unresectable, malignant obstruction where ERCP fails: endoscopic ultrasonography-guided choledochoduodenostomy versus percutaneous drainage. J Clin Gastroenterol. 2012 Oct;46(9):768-74. doi: 10.1097/MCG.0b013e31825f264c. PMID 22810111
- [Background] Khashab MA, Valeshabad AK, Afghani E, Singh VK, Kumbhari V, Messallam A, Saxena P, El Zein M, Lennon AM, Canto MI, Kalloo AN. A comparative evaluation of EUS-guided biliary drainage and percutaneous drainage in patients with distal malignant biliary obstruction and failed ERCP. Dig Dis Sci. 2015 Feb;60(2):557-65. doi: 10.1007/s10620-014-3300-6. Epub 2014 Aug 1. PMID 25081224
- [Background] Sharaiha RZ, Kumta NA, Desai AP, DeFilippis EM, Gabr M, Sarkisian AM, Salgado S, Millman J, Benvenuto A, Cohen M, Tyberg A, Gaidhane M, Kahaleh M. Endoscopic ultrasound-guided biliary drainage versus percutaneous transhepatic biliary drainage: predictors of successful outcome in patients who fail endoscopic retrograde cholangiopancreatography. Surg Endosc. 2016 Dec;30(12):5500-5505. doi: 10.1007/s00464-016-4913-y. Epub 2016 Apr 29. PMID 27129552
- [Background] Lee TH, Choi JH, Park do H, Song TJ, Kim DU, Paik WH, Hwangbo Y, Lee SS, Seo DW, Lee SK, Kim MH. Similar Efficacies of Endoscopic Ultrasound-guided Transmural and Percutaneous Drainage for Malignant Distal Biliary Obstruction. Clin Gastroenterol Hepatol. 2016 Jul;14(7):1011-1019.e3. doi: 10.1016/j.cgh.2015.12.032. Epub 2015 Dec 31. PMID 26748220
- [Background] Sportes A, Camus M, Greget M, Leblanc S, Coriat R, Hochberger J, Chaussade S, Grabar S, Prat F. Endoscopic ultrasound-guided hepaticogastrostomy versus percutaneous transhepatic drainage for malignant biliary obstruction after failed endoscopic retrograde cholangiopancreatography: a retrospective expertise-based study from two centers. Therap Adv Gastroenterol. 2017 Jun;10(6):483-493. doi: 10.1177/1756283X17702096. Epub 2017 Apr 10. PMID 28567118
- [Background] Schmitz D, Grosse A, Hallscheidt P, Roseneck A, Niemeyer J, Rudi J. Color Doppler ultrasound-guided PTBD with and without metal stent implantation by endoscopic control: prospective success and early adverse event rates. Z Gastroenterol. 2015 Nov;53(11):1255-60. doi: 10.1055/s-0041-104225. Epub 2015 Nov 12. PMID 26562399
- [Background] Liu YS, Lin CY, Chuang MT, Tsai YS, Wang CK, Ou MC. Success and complications of percutaneous transhepatic biliary drainage are influenced by liver entry segment and level of catheter placement. Abdom Radiol (NY). 2018 Mar;43(3):713-722. doi: 10.1007/s00261-017-1258-5. PMID 28741168
- [Derived] Schmitz D, Valiente CT, Dollhopf M, Perez-Miranda M, Kullmer A, Gornals J, Vila J, Weigt J, Voigtlander T, Redondo-Cerezo E, von Hahn T, Albert J, Vom Dahl S, Beyna T, Hartmann D, Franck F, Garcia-Alonso FJ, Schmidt A, Garcia-Sumalla A, Arrubla A, Joerdens M, Kleemann T, Tomo JRA, Grassmann F, Rudi J. Percutaneous transhepatic or endoscopic ultrasound-guided biliary drainage in malignant distal bile duct obstruction using a self-expanding metal stent: Study protocol for a prospective European multicenter trial (PUMa trial). PLoS One. 2022 Oct 27;17(10):e0275029. doi: 10.1371/journal.pone.0275029. eCollection 2022. PMID 36302047